CLINICAL TRIAL: NCT05824858
Title: A Phase 1 Study to Evaluate the Effect of Food on the LY3537982 Pharmacokinetics in Health Adult Subjects
Brief Title: A Study of the Effect of Food on LY3537982 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-RAS-23006; J3M-OX-JZQI (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3537982 (High-Fat Meal) (Experimental): LY3537982 administered orally under fasting conditions in one study period and under fed conditions (i.e., a standard high-fat meal) in the other study period.
  Interventions: Drug: LY3537982
- LY3537982 (Low-Fat Meal) (Experimental): LY3537982 administered orally under fasting conditions in one study period and under fed conditions (i.e., a standard low-fat meal) in the other study period.
  Interventions: Drug: LY3537982

INTERVENTIONS:
Drug: LY3537982 — Administered orally.

SUMMARY:
The main purpose of this study is to conduct blood tests to measure how much LY3537982 is in the bloodstream and how the body handles and eliminates LY3537982 after meals and on an empty stomach. The study will also evaluate the safety and tolerability of LY3537982. Participants will stay in the research center during the study, which will last about one week, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Healthy status as defined by the absence of evidence of any clinically significant active or chronic disease
* Body mass index (BMI): 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive

Exclusion Criteria:

* Females who are lactating or of childbearing potential
* Clinically significant history of any drug sensitivity, drug allergy, or food allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-06-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration-Time Curve (AUC) from Time 0 to Infinity (AUC[0-inf]) | Day 1 and Day 4 of each study period
  PK: AUC(0-inf)
PK: Maximum Observed Concentration (Cmax) of LY3537982 | Day 1 and Day 4 of each study period
  PK: Cmax of LY3537982

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Guo-Avrutin, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- ICON, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No